CLINICAL TRIAL: NCT00170677
Title: Topotecan Weekly Versus Topotecan Day 1-5 in Patient With Platin-resistant Ovarian Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: North Eastern German Society of Gynaecological Oncology (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 4401000
Record Dates: First submitted 2005-09-13; First posted 2005-09-15 (Estimated); Last update posted 2014-05-14 (Estimated); Status verified 2010-07

CONDITIONS: Ovarian Cancer
MeSH Terms: conditions — Ovarian Neoplasms | interventions — Topotecan

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- A (Active Comparator)
  Interventions: Drug: Topotecan
- B (Experimental)
  Interventions: Drug: Topotecan

INTERVENTIONS:
Drug: Topotecan — Topotecan 4,0 mg/m² administered in day 1, 8 und 15 as i.v. infusion for 30 minutes. A cycle lasts 28 days.
  Arms: B
Drug: Topotecan — Topotecan 1,25 mg/m²/day, day 1-5 as i.v. infusion of 30 minutes. Repeat after 21 day.
  Arms: A

SUMMARY:
Comparison of topotecan weekly vs. topotecan day 1-5. The compatibility and activity are to be examined.

DETAILED DESCRIPTION:
Topotecan belongs to the most effective medicaments in the therapy of relapsed platin-resistant ovarian cancer. Due to the low rate of hematological toxicities of grade 3 or 4 weekly application may be an improvement of therapy. None randomised study exists comparing a weekly topotecan application with an application on day 1-5. This study will compare the two applications in regard to: rate of complete or partial remissions, rate of toxicity, quality of life, progression free survival, overall survival.

ELIGIBILITY:
Inclusion Criteria:

* patients with histologically-confirmed ovarian cancer
* relapse within 6 month after primary therapy
* primary therapy with platin and taxan
* ECOG 0-2
* >= 18 years
* leukocytes >= 3.000/ µl
* platelet >= 100.000/ µl
* neutrophil >= 1.500/ µl
* written informed consent

Exclusion Criteria:

* earlier topotecan therapy
* simultaneous or planned radiotherapy
* secondary malignancy

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 194 (Actual)
Dates: Start 2005-09; Primary Completion 2013-01 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
Rate of CR and PR in each arm | every 12 weeks

SECONDARY OUTCOMES:
Toxicity of topotecan treatment | after each cycle
Progression-free survival of both arms | every 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Werner Lichtenegger, Study Chair — Charite University, Berlin, Germany
Locations (1):
- Charité Campus Virchow-Klinikum, Berlin, Germany